CLINICAL TRIAL: NCT04568083
Title: An Observational, Register-based Study on Ticagrelor 60 mg Persistence and Event Rates in Clinical Practice in the US and Europe.
Brief Title: Patient Characteristics, Persistence to Treatment and Outcome Events in Patients Treated With Ticagrelor 60 mg After Myocardial Infarction in Real-world Clinical Practice
Acronym: ALETHEIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130R00057
Record Dates: First submitted 2020-09-15; First posted 2020-09-29 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Infarction (MI)
Keywords: Myocardial Infarction; Ticagrelor 60 mg; Antiplatelet agents; Medication persistence; Drug utilization; Bleeding; MACE; Cardiovascular; Cohort study; Observational study; Real-world evidence
MeSH Terms: conditions — Myocardial Infarction; Medication Adherence; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ticagrelor cohort: Patients initiating ticagrelor 60 mg after an MI, with no prescription of ticagrelor 60 mg prior to their qualifying MI. The qualifying MI is defined as the most recent MI occurring before the first ticagrelor 60 mg prescription.
- Non-ticagrelor cohort: Patients not prescribed ticagrelor 60 mg at a comparable time point after an MI as matched patients in the ticagrelor cohort. Patients may be prescribed another P2Y12 inhibitor or aspirin alone.

SUMMARY:
This is an observational study based on secondary data extracted from multiple register-based data sources in the US and Europe (Sweden, United Kingdom, Italy, Germany). The study will include patients initiating treatment with ticagrelor 60 mg after a myocardial infarction in real-world clinical practice, and describe their patient characteristics and duration of treatment. If the a priori threshold of 5,000 person-years on treatment with ticagrelor 60 mg is met, outcome events (bleeding and cardiovascular events) will also be analysed and described.

DETAILED DESCRIPTION:
This observational cohort study will include patients initiating treatment with ticagrelor 60 mg after a myocardial infarction (MI), and describe their patient characteristics and persistence to treatment. To contextualise the characteristics of the ticagrelor patients, two reference cohorts will be created, including patients treated with another P2Y12 inhibitor than ticagrelor (clopidogrel, prasugrel, or ticlopidine), and patients not treated with any P2Y12 inhibitor, within a comparable timepoint from an MI as for the ticagrelor 60 mg patients. If the a priori threshold of 5,000 person-years on treatment with ticagrelor 60 mg is met, to ensure sufficient precision, outcome events (bleeding and cardiovascular events) will also be analysed and described. Outcome events will only be described in the ticagrelor cohorts; no comparison of outcomes will be made between the ticagrelor and the reference cohorts.

The primary outcome is bleeding requiring hospitalisation. The secondary outcomes include components of the primary outcome, and cardiovascular outcomes. Persistence to treatment with ticagrelor 60 mg will also be assessed The study will be performed in the US and 4 European countries (Sweden, United Kingdom, Italy, Germany).

ELIGIBILITY:
Inclusion Criteria:

Primary Analysis Population:

* Hospitalisation with a primary diagnosis of MI during the eligibility period
* Ticagrelor cohort: A first prescription of ticagrelor 60 mg after the most recent hospitalisation with a primary diagnosis of MI.
* Non-ticagrelor cohort: A prescription of clopidogrel, prasugrel or ticlopidine, or no prescription for any of these medications, at a comparable timepoint relative to their MI as for the ticagrelor cohort

Secondary Analysis Population:

* The qualifying prescription 12-36 months after a hospitalisation with a primary diagnosis of MI and treatment with an ADP receptor antagonist (clopidogrel, prasugrel, ticagrelor 90 mg, ticlopidine) ≤12 months prior to the qualifying prescription, or the qualifying prescription 12-24 months after a hospitalisation with a primary diagnosis of MI AND
* Age ≥50 years
* At least one of the following risk factors:

  * Age ≥ 65 years
  * Diabetes mellitus requiring medication
  * A second prior MI
  * Evidence of multivessel coronary artery disease
  * Chronic non-end-stage renal dysfunction

Exclusion Criteria:

Applicable to the Primary and Seconday Analysis Populations:

* Dies, emigrates, or disenrolls from the database (where applicable) prior to the ticagrelor approval date.
* Ineligibility for ticagrelor use (restricted to the conditions possible to capture within the data sources)-one or more of the following:

  * Concomitant use of an anticoagulant
  * Prior ischaemic stroke
  * Prior history of intracranial bleeding
  * Severe hepatic impairment
  * Gastrointestinal bleeding
  * Renal failure requiring dialysis
  * Concomitant use of a strong CYP3A4 inhibitor or inducer
* <1 year of data available prior to the qualifying MI (for assessment of patient characteristics at qualifying MI)

Max Age: 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients who are hospitalised with a primary diagnosis of MI, identified using diagnostic codes, divided into cohorts receiving and not receiving treatment with ticagrelor 60 mg. Co-prescription of aspirin will also be identified where available.
Sampling Method: Non-Probability Sample
Enrollment: 7035 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Treatment persistence | From initiation of ticagrelor 60 mg to discontinuation, switch or death, assessed throughout the study period up to a maximum of 36 months
  Treatment discontinuation is defined on the basis of calculated days of supply from prescription data.
Incidence of Major bleeding | From initiation of ticagrelor 60 mg until the date of a major bleeding event, assessed throughout the study period until treatment discontinuation or end of follow-up, up to a maximum of 36 months
  Major bleeding is defined as bleeding requiring hospitalisation.

SECONDARY OUTCOMES:
Incidence of Bleeding events | From initiation of ticagrelor 60 mg until the date of a bleeding event, assessed throughout the study period until treatment discontinuation or end of follow-up, up to a maximum of 36 months
  * Intracranial haemorrhage
  * Gastrointestinal bleeding requiring hospitalisation
  * Bleeding other than intracranial haemorrhage or gastrointestinal bleeding requiring hospitalisation
  * Fatal bleeding
  * Bleeding not requiring hospitalisation (managed in outpatient care/emergency care not requiring hospitalisation)
Incidence of Cardiovascular (CV) events | From initiation of ticagrelor 60 mg until the date of a CV event, assessed throughout the study period until treatment discontinuation or end of follow-up, up to a maximum of 36 months
  * Composite of hospitalisation for MI or stroke, and all-cause mortality
  * Composite of hospitalisation for MI or stroke, and CV death (three-point MACE)
  * Hospitalisation for MI, hospitalisation for stroke, hospitalisation for ischaemic stroke, CV death, CHD death, all-cause mortality assessed individually

OTHER OUTCOMES:
Incidence of Dyspnoea | From initiation of ticagrelor 60 mg until the date of a dyspnoea event, assessed throughout the study period until treatment discontinuation or end of follow-up, up to a maximum of 36 months
  Dyspnoea is assessed as dyspnoea diagnosed in any setting, as well as dyspnoea requiring hospitalisation, where data availability allows.
Incidence of Amputation (lower-limb) | From initiation of ticagrelor 60 mg until the date of amputation of lower limb, assessed throughout the study period until treatment discontinuation or end of follow-up, up to a maximum of 36 months
  Amputation (lower-limb) is defined as hospitalisation with a procedure code for amputation of lower limb.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Research Site, Bethesda, Maryland
  - Research Site, Waltham, Massachusetts
- Research Site, Wismar, Germany
- Research Site, Rome, Italy
- Research Site, Stockholm, Sweden
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bonaca MP, Lesen E, Giannitsis E, Hedberg J, Jernberg T, Lambrelli D, Duong M, Maggioni AP, Ariza-Sole A, Ten Berg J, Storey RF. Characteristics and outcomes in patients with a prior myocardial infarction treated with extended dual antiplatelet therapy with ticagrelor 60 mg: findings from ALETHEIA, a multi-country observational study. Eur Heart J Cardiovasc Pharmacother. 2023 Dec 14;9(8):701-708. doi: 10.1093/ehjcvp/pvad062. PMID 37653447
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5130R00057&attachmentIdentifier=a94f5caf-f7fb-4b22-903e-05a05af84939&fileName=D5130R00057_ALETHEIA_CSR_Synopsis.pdf&versionIdentifier=